CLINICAL TRIAL: NCT02641236
Title: A Randomized Phase 2 Study to Examine the Impact of Gut Decontamination on Intestinal Microbiome Composition in Pediatric Allogeneic Hematopoietic Stem Cell Transplant Patients
Brief Title: Gut Decontamination In Pediatric Allogeneic Hematopoietic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Leslie Lehmann, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-394
Record Dates: First submitted 2015-11-16; First posted 2015-12-29 (Estimated); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Hematopoietic Stem Cell Transplantation (HSCT); Acute GVH Disease
Keywords: Hematopoietic Stem Cell Transplantation (HSCT); Acute GVH Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gut Decontamination with vancopoly (Active Comparator): * All eligible participants will be randomized to either Arm A: "Gut Decontamination" or Arm B: "No Gut Decontamination".
  * Participants assigned to this arm will receive non-absorbable, oral vancomycin-polymyxin B as per our institutional standard practice.
  Interventions: Drug: Vancomycin-polymyxin B
- No Gut Decontamination (No Intervention): * All eligible participants will be randomized to either Arm A: "Gut Decontamination" or Arm B: "No Gut Decontamination".
  * Participants assigned to this arm will not receive oral vancomycin-polymyxin B, but all other HSCT supportive care will be the same as for patients in Arm A.

INTERVENTIONS:
Drug: Vancomycin-polymyxin B
  Arms: Gut Decontamination with vancopoly

SUMMARY:
This research study is for participants who are undergoing allogeneic hematopoietic stem cell transplantation (HSCT) and are at risk for developing acute graft-versus-host disease (GVHD). GVHD is a complication of HSCT in which immune cells from the donor cause inflammation and injury to tissues and organs of the HSCT recipient. Vancomycin-polymyxin B (commonly called "vancopoly") is an oral antibiotic that is given to people undergoing allogeneic HSCT as a preventive measure for acute GVHD. This research study is studying the effects of vancopoly on the microorganisms living in the intestine during and after stem cell transplantation.

DETAILED DESCRIPTION:
This research study is a Phase 2 clinical trial. Phase 2 clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease.

"Investigational" means that the intervention is being studied.

Pre-clinical studies performed in the 1970's showed that killing all the bacteria in the intestine with oral antibiotics could decrease the risk of acute GVHD following allogeneic HSCT. Based on this observation, many stem cell transplant centers adopted the practice of "gut decontamination" with oral antibiotics as a preventive measure for acute GVHD. There is no standard regimen for gut decontamination between transplant centers, and there are no definitive human studies showing that gut decontamination is beneficial for lowering the risk of acute GVHD.

Recent studies in adult patients undergoing stem cell transplant indicate that the types of bacteria living in the intestine can influence bone marrow transplant outcomes such as survival and development of acute GVHD. Some types of bacteria may be protective against GVHD and others may increase the risk of GVHD. Based on this newer research, it is possible that the practice of gut decontamination ("vancopolys") may not be beneficial for HSCT patients.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility Criteria for Patients Undergoing Allogeneic HSCT

  * Recipient of 9/10 or 10/10 (HLA-A, -B, -C, -DRB1, -DQB1) matched bone marrow allogeneic hematopoietic stem cell transplantation (HSCT) OR 4/6, 5/6 and 6/6 (HLA-A, -B, -DR) matched cord blood allogeneic HSCT.
  * Participants may have underlying malignant or non-malignant hematologic disease, except for primary immunodeficiency, as the indication for their allogeneic HSCT. Patients with immune dysregulation such as familial or secondary hemophagocytic lymphohistiocytosis (HLH) are eligible.
  * Participants must may receive either a myeloablative or non-myeloablative(reduced-intensity) conditioning regimen. Anti-thymocyte globulin (ATG) in the conditioning regimen is permitted.
  * Graft-versus-host disease (GVHD) prophylaxis with any of the following agents: calcineurin inhibitor, and short-course methotrexate, with or without steroids, mycophenolate mofetil, and sirolimus.
  * Age ≥ 4 years old and toilet-trained. Participants must be able to deposit stool samples directly into stool collection containers. Stool specimens from diapers are difficult to obtain and are prone to more sampling error, particularly for loose or liquid stools which are common in the peri-transplant period.
  * Lansky/Karnofsky performance status ≥60% (see Appendix A)
  * Ability to understand and/or the willingness of their parent or legally authorized representative to sign a written informed consent document
* Eligibility Criteria for Healthy Bone Marrow Donors

  * Healthy individuals, ages ≥ 4 years and toilet-trained, who have been identified by BCH or DFCI providers as 9/10 or 10/10 (HLA-A, -B, -C, -DRB1, -DQB1 matched bone marrow donors for transplantation will also be eligible to participate in this study.

Exclusion Criteria:

* Patients undergoing allogeneic HSCT for correction of a primary immunodeficiency disorder (e.g. SCID).
* Patients with age ≤ 10 years undergoing HSCT with a matched sibling donor. These patients are at very low risk of acute GVHD and do not receive gut decontamination per our institutional standard practice.
* Participants receiving GVHD prophylaxis with drugs other than calcineurin inhibitors, methotrexate or steroids.agents listed above (e.g. abatacept).
* History of allergic reactions attributed to oral vancomycin or oral polymyxin B.
* Participants undergoing active therapy for immune-mediated or infectious colitis upon admission for allogeneic HSCT.
* Participants receiving antibiotic therapy for treatment of a bacterial infection or bacterial prophylaxis upon admission for allogeneic HSCT. Use of any agent (e.g. sulfamethoxazole/trimethoprim) for prophylaxis of Pneumocystis jirovecii pneumonia is permitted. Concurrent use of anti-fungal and anti-viral therapies is also permitted.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 4 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03; Primary Completion 2021-04-15 (Actual); Study Completion 2021-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Lehmann, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Severyn CJ, Siranosian BA, Kong ST, Moreno A, Li MM, Chen N, Duncan CN, Margossian SP, Lehmann LE, Sun S, Andermann TM, Birbrayer O, Silverstein S, Reynolds CG, Kim S, Banaei N, Ritz J, Fodor AA, London WB, Bhatt AS, Whangbo JS. Microbiota dynamics in a randomized trial of gut decontamination during allogeneic hematopoietic cell transplantation. JCI Insight. 2022 Apr 8;7(7):e154344. doi: 10.1172/jci.insight.154344. PMID 35239511

RESULTS

PARTICIPANT FLOW:
Groups:
- Gut Decontamination With Vancopoly: * All eligible participants will be randomized to either Arm A: "Gut Decontamination" or Arm B: "No Gut Decontamination".
  * Participants assigned to this arm will receive non-absorbable, oral vancomycin-polymyxin B starting on Day -5, relative to stem cell infusion (Day 0) and continue through neutrophil engraftment.
  Vancomycin-polymyxin B dosing is based off of body surface area (bsa):
  * Subjects with a bsa < 0.5 m2 will take 1 capsule, administered orally (PO), three times a day (TID).
  * Subjects with a bsa of 0.5-0.99 m2 will take 2 capsules, PO, TID.
  * Subjects with a bsa of 1-1.49 m2 will take 3 capsules, PO, TID.
  * Subjects with a bsa > or =1.5 m2 will take 4 capsules, PO, TID.
- Healthy Donor Control Group: Eligible subjects will be registered to the study. Healthy donors will not receive any treatment on the study. Healthy donors will provide a stool sample around the time of the donor evaluation visit or donor bone marrow harvest. Additional stool samples may be collected at the 6 months post-transplant and 1 year post-transplant timepoints. Donor stool samples will be compared to their corresponding recipient's stool samples. Additionally, healthy donors will provide a one time peripheral blood sample at the time of the evaluation visit or donor bone marrow harvest. The volume of blood will not exceed 30ml or 3ml/kg, whichever is less.
Period: Overall Study
Arm/Group | Gut Decontamination With Vancopoly | No Gut Decontamination | Healthy Donor Control Group
Started | 10 | 10 | 4
Completed | 5 | 3 | 4
Not Completed | 5 | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Gut Decontamination With Vancopoly: * All eligible participants will be randomized to either Arm A: "Gut Decontamination" or Arm B: "No Gut Decontamination".
  * Participants assigned to this arm will receive non-absorbable, oral vancomycin-polymyxin B as per our institutional standard practice.
  Vancomycin-polymyxin B
- Healthy Donor Control Group: -Healthy individuals, ages 4 years old and older and toilet trained, who have been identified as 9/10 or 10/10 matched, bone marrow donors for transplantation. Healthy donors may be related or unrelated to the bone marrow recipient.
- Total: Total of all reporting groups
Arm/Group | Gut Decontamination With Vancopoly | No Gut Decontamination | Healthy Donor Control Group | Total
Number analyzed (Participants) | 10 | 10 | 4 | 24
Age, Customized [Mean (Full Range); unit: years] — Population: Healthy donor control group did not receive transplant, so 'Age at Transplant' were not capable to be collected for this group.
  years
    Age at transplant: number analyzed (Participants) | 10 | 10 | 0 | 20
    Age at transplant | 13.4 [8 to 24.4] | 18.7 [7.1 to 24.6] |  | 15.2 [7.1 to 24.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 2 | 12
  Male | 3 | 7 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 0 | 6
  Not Hispanic or Latino | 5 | 8 | 4 | 17
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 10 | 4 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Primary disease [Count of Participants; unit: Participants] — Population: Healthy Donor Control Group subjects do not have a Primary Disease.
  Participants
    number analyzed (Participants) | 10 | 10 | 0 | 20
    Acute lymphocytic leukemia (ALL) | 4 | 4 | 0 | 8
    Acute myeloid leukemia (AML) | 1 | 4 | 0 | 5
    Myelodysplastic syndromes (MDS) | 2 | 0 | 0 | 2
    Anemia/red blood cell disorder | 3 | 2 | 0 | 5
Conditioning regimen intensity [Count of Participants; unit: Participants] — Population: Healthy Donor Control subjects did not receive transplants.
  Participants
    number analyzed (Participants) | 10 | 10 | 0 | 20
    Myeloablative | 8 | 9 | 0 | 17
    Nonmyeloablative | 2 | 1 | 0 | 3
Human leukocyte antigen (HLA) molecular typing [Count of Participants; unit: Participants] — Human leukocyte antigen (HLA) molecular typing is run through the American Red Cross (ARC). HLA typing is performed by polymerase chain reaction sequence-specific oligonucleotide probes, Sanger sequence based typing, and next generation sequencing. Transplant recipients will have one high resolution result and one result from a buccal swab sample performed by the ARC. Both samples are processed using the same methods. Typing was performed at 5 loci (HLA-A, -B, -C, -DRB1, and -DQB1). Fully HLA-matched is considered a 10/10 match at all 5 loci, and a 9/10 match was considered HLA-mismatched. Population: Data not collected from Healthy Donor Control Group.
  Participants
    number analyzed (Participants) | 10 | 10 | 0 | 20
    Matched related | 5 | 1 | 0 | 6
    Mismatch related | 0 | 1 | 0 | 1
    Matched unrelated | 2 | 5 | 0 | 7
    Mismatch unrelated | 3 | 3 | 0 | 6
Patient or donor serostatus [Count of Participants; unit: Participants] — Population: Data not collected from Healthy Donor Control Group.
  Participants
    number analyzed (Participants) | 10 | 10 | 0 | 20
    Positive | 5 | 8 | 0 | 13
    Negative | 5 | 2 | 0 | 7
Patient/donor sex mismatch [Count of Participants; unit: Participants] — Population: Data not collected from Healthy Donor Control Group.
  Participants
    number analyzed (Participants) | 10 | 10 | 0 | 20
    F to M | 2 | 2 | 0 | 4
    Other | 8 | 8 | 0 | 16
Graft source [Count of Participants; unit: Participants] — Population: Healthy Donor Control subjects did not receive transplants.
  Participants
    number analyzed (Participants) | 10 | 10 | 0 | 20
    Bone marrow | 9 | 10 | 0 | 19
    Cord | 1 | 0 | 0 | 1
Graft Versus Host Disease (GVHD) prophylaxis [Count of Participants; unit: Participants] — Population: Healthy Donor Control subjects did not receive transplants.
  Participants
    number analyzed (Participants) | 10 | 10 | 0 | 20
    Cyclosporine (CsA) | 1 | 0 | 0 | 1
    CsA/ Methotrexate (MTX) +/- methylprednisone | 8 | 9 | 0 | 17
    CsA/ Mycophenolate mofetil (MMF) | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Gut Microbiome Description
Description: Shannon diversity index (range: 0-6), measured at 2 weeks post stem cell transplant. Shannon diversity is a way to calculate biodiversity in a community, and assumes that all species are represented in a sample and that they are randomly sampled. Shannon Diversity is a measurement sensitive to the loss of rare taxa (34 in the JCI Insight manuscript, Konopinski MK, PeerJ. 2020;8:e9391) and estimates microbial richness (e.g., the number of species) and evenness (e.g., the relative abundance of organisms within a sample).
  Formula 1: H = -∑[(pi) * ln(pi)],
  * H: Shannon diversity index (H = 0 indicates that a community has only one species) pi: Proportion of individuals of i-th species in a whole community Formula 2: pi = n / N,
  * n: individuals of a given type/species
  * N: total number of individuals in a community
Time Frame: 2 Weeks post HSCT
Measure: Median (Full Range); unit: Shannon diversity index
Arm/Group | Gut Decontamination With Vancopoly | No Gut Decontamination
Number analyzed (Participants) | 10 | 10
Shannon diversity index | 2.4 [0.03 to 5.32] | 3.1 [2.1 to 3.7]

2. Secondary Outcome: Diarrhea Frequency
Description: The number of daily bowel movements during the first 7 days post-HSCT is charted by floor nurses and/or clinical assistants and will be obtained from within each patient's electronic medical record in PowerChart. Diarrhea frequency is defined the proportion of participants who had greater than 3 bowel movements per day.
Time Frame: Participants were followed 7 days after HSCT.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Gut Decontamination With Vancopoly | No Gut Decontamination
Number analyzed (Participants) | 10 | 10
proportion of participants | 0.4 [0.15 to 0.70] | 0.4 [0.15 to 0.70]

3. Secondary Outcome: Median Absolute Cell Numbers of T-, B-, NK- and Dendritic Cell Subsets by Flow Cytometry
Description: CD4+ Tregs were defined as CD3+CD4+CD25med-hiCD127lo, CD4+; Tcon as CD3+CD4+CD25neg-lo CD127med-hi, B cells as CD19+, cytotoxic T cells as CD8+, and natural killer cells as CD56+CD3-. Within CD4+ Tregs and CD4+ Tcon, subsets were defined as follows: naive T cells (CD45RO-CD62L+), central memory (CD45RO+CD62L+), and effector memory (CD45RO+CD62L-).
Time Frame: Performed at the post-transplant time points (1,2,3,6,9,12 months post-transplant)
Population: Excluding two patients with graft failure.
Measure: Median (Full Range); unit: number of cells per microliter
Arm/Group | Gut Decontamination With Vancopoly | No Gut Decontamination
Number analyzed (Participants) | 9 | 9
number of cells per microliter
  CD4+ at 1 month | 80.95 [3.72 to 195.49] | 119.78 [5.99 to 725.56]
  CD4+ at 2 months | 99.89 [59.01 to 190.76] | 81.92 [8.31 to 285.83]
  CD4+ at 3 months | 126.54 [23.72 to 246.35] | 182.09 [9.97 to 312.63]
  CD4+ at 6 months | 206.50 [123.18 to 675.64] | 248.24 [44.29 to 739.08]
  CD4+ at 9 months | 230.28 [161.54 to 565.65] | 335.43 [37.39 to 458.98]
  CD4+ at 12 months | 380.22 [200.19 to 459.49] | 429.53 [6.74 to 524.61]
  Treg/Tcon at 1 month | 0.10 [0.04 to 0.55] | 0.12 [0.06 to 0.43]
  Treg/Tcon at 2 months | 0.10 [0.02 to 0.43] | 0.12 [0.01 to 0.14]
  Treg/Tcon at at 3 months | 0.091 [0.021 to 0.255] | 0.098 [0.013 to 0.130]
  Treg/Tcon at 6 months | 0.088 [0.020 to 0.295] | 0.098 [0.043 to 0.181]
  Treg/Tcon at at 9 months | 0.094 [0.062 to 0.176] | 0.072 [0.035 to 0.218]
  Treg/Tcon at 12 months | 0.080 [0.071 to 0.298] | 0.088 [0.046 to 0.115]
  CD8+ at 1 month | 126.44 [3.56 to 408.70] | 39.40 [3.06 to 751.53]
  CD8+ at 2 months | 89.12 [53.44 to 681.27] | 111.19 [36.31 to 1191.26]
  CD8+ at 3 months | 401.16 [20.64 to 1432.25] | 191.32 [13.90 to 1158.49]
  CD8+ at 6 months | 331.87 [63.76 to 820.64] | 270.11 [93.85 to 2895.98]
  CD8+ at 9 months | 302.13 [137.93 to 455.02] | 206.93 [40.67 to 3131.85]
  CD8+ at 12 months | 317.51 [182.15 to 618.93] | 394.30 [11.64 to 2919.11]
  CD4+ Tcon naive at 1 month | 0.08 [0.00 to 0.44] | 0.04 [0.01 to 0.57]
  CD4+ Tcon naive at 2 months | 0.17 [0.04 to 0.35] | 0.02 [0.003 to 0.18]
  CD4+ Tcon naive at 3 months | 0.09 [0.02 to 0.42] | 0.05 [0.02 to 0.26]
  CD4+ Tcon naive at 6 months | 0.11 [0.04 to 0.70] | 0.11 [0.002 to 0.33]
  CD4+ Tcon naive at 9 months | 0.32 [0.09 to 0.86] | 0.05 [0.02 to 0.57]
  CD4+ Tcon naive at 12 months | 0.41 [0.37 to 0.54] | 0.31 [0.05 to 0.61]
  B-cells at 1 month | 2.06 [0.00 to 25.02] | 2.75 [0.55 to 55.25]
  B-cells at 2 months | 14.26 [0.00 to 84.63] | 1.85 [0.77 to 258.41]
  B-cells at 3 months | 60.39 [1.94 to 161.10] | 8.07 [0.55 to 126.58]
  B-cells at 6 months | 261.38 [29.75 to 418.49] | 103.25 [1.43 to 199.00]
  B-cells at 9 months | 617.48 [0.81 to 928.48] | 250.69 [1.83 to 357.38]
  B-cells at 12 months | 903.44 [579.11 to 1195.48] | 223.92 [0.04 to 460.35]
  NK cells at 1 month | 46.92 [5.39 to 406.13] | 79.89 [23.28 to 1264.25]
  NK cells at 2 months | 104.42 [57.68 to 270.51] | 123.61 [14.07 to 295.87]
  NK cells at 3 months | 109.50 [20.43 to 276.17] | 136.75 [26.35 to 230.76]
  NK cells at 6 months | 209.84 [117.32 to 346.88] | 111.80 [36.17 to 293.05]
  NK cells at 9 months | 187.37 [32.95 to 333.75] | 137.90 [61.41 to 239.08]
  NK cells at 12 months | 193.19 [37.87 to 338.91] | 100.42 [9.86 to 215.03]

4. Secondary Outcome: Incidence of Acute GVHD (Grade 2-4)
Description: Grade 2 acute GVHD was defined as skin stage 3 or GI stage 1 or liver stage 1. Skin stage 3 was defined as maculopapular rash >50% of body surface or generalized erythroderma; GI stage 1 was defined as adults: 500 - 1000 mL/day, children: 10 - 19.9 mL/kg/day or nausea, anorexia or vomiting with biopsy (EGD) confirmation of upper GI GVHD; liver stage 1 was defined as bilirubin 2.1-3 mg/dL. Grade 3 acute GVHD was defined as GI stage 2-4 or liver stage 2-3. GI stage 2-4 was defined as >1001 mL/day (adults), >30 ml/kg/day(children) or large volume stool with severe abdominal pain with our whiteout ileus or stool with frank blook or melena; liver stage 2-3 was defined as bilirubin 3.1-15mg/dL. Grade 4 acute GVHD was defined as skin stage 4 or liver stage 4. Skin stage 4 was defined as generalized erythroderma with bullous formation and desquamation; liver stage 4 was defined as bilirubin > 15mg/dL.
Time Frame: Each stool collection time point after neutrophil engraftment until day +100
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Gut Decontamination With Vancopoly | No Gut Decontamination
Number analyzed (Participants) | 10 | 10
proportion of participants
  Grade 2 | 0.10 [0.003 to 0.45] | 0 [0 to 0.31]
  Grade 3-4 | 0 [0 to 0.31] | 0.30 [0.07 to 0.65]

5. Secondary Outcome: Overall Survival Rate at 12 Months (OS12)
Description: OS12 is the proportion of participants alive at 12 months after study entry.
Time Frame: All participants were followed for 1 years after study entry.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Gut Decontamination With Vancopoly | No Gut Decontamination
Number analyzed (Participants) | 10 | 10
proportion of participants | 1 [0.69 to 1] | 1 [0.69 to 1]

6. Secondary Outcome: Relapse Free Rate at 12 Months
Description: Relapse free rate at 12 months was defined as the proportion of patients surviving without any signs or symptoms of that cancer after 12 months.
Time Frame: Patients were followed for 12 months.
Population: The analysis is comprised of participants with a malignancy.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Gut Decontamination With Vancopoly | No Gut Decontamination
Number analyzed (Participants) | 7 | 8
proportion of participants | 0.57 [0.18 to 0.90] | 0.75 [0.35 to 0.97]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of consent until the subject reached 24 months post-transplant or until they were taken off study, whichever came first. Subjects in the Healthy Donor Control Group were not monitored/ for Adverse Events.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv4. All remaining events regardless of treatment attribution were classified as Other AEs. Per the source vocabulary (CTCAEv4.0) there is a category "Other, specify" for each system organ class. No further data is available to specify classification beyond this general term.
Arm/Group | Gut Decontamination With Vancopoly | No Gut Decontamination | Healthy Donor Control Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/10 | 3/10 | 0/0
Other Adverse Events (participants affected / at risk) | 8/10 | 2/10 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gut Decontamination With Vancopoly (N=10) | No Gut Decontamination (N=10) | Healthy Donor Control Group (N=0)
Blood Bilirubin Increased (Blood and lymphatic system disorders) | 0 | 1 | NA
ALT Increase (Blood and lymphatic system disorders) | 1 | 2 | NA
AST Increased (Blood and lymphatic system disorders) | 1 | 1 | NA
Hepatobiliary disorders (Hepatobiliary disorders) | 1 | 0 | NA — Hepatobiliary disorders, other - VOD
Hypotension (Cardiac disorders) | 1 | 0 | NA
Hypokalemia (Blood and lymphatic system disorders) | 1 | 0 | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | NA
GGT Increased (Blood and lymphatic system disorders) | 0 | 1 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gut Decontamination With Vancopoly (N=10) | No Gut Decontamination (N=10) | Healthy Donor Control Group (N=0)
Mucositis (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Abdominal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acidosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 0 | 0
ALT Increased (Blood and lymphatic system disorders) | 3 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 0
AST Increased (Blood and lymphatic system disorders) | 2 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Blood Bilirubin Increased (Blood and lymphatic system disorders) | 3 | 0 | 0
Creatinine Increased (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 | 1 | 0
Upper GI GVHD (Gastrointestinal disorders) | 1 | 0 | 0
Hepatobiliary disorder, other- VOD (Hepatobiliary disorders) | 1 | 0 | 0
Hypernatremia (Blood and lymphatic system disorders) | 1 | 0 | 0
Hypertension (Cardiac disorders) | 4 | 0 | 0
Hypokalemia (Blood and lymphatic system disorders) | 4 | 0 | 0
Hypophosphatemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Hypotension (Cardiac disorders) | 1 | 0 | 0
Hypoxia (Vascular disorders) | 5 | 0 | 0
Infections and infestations, other- CMV reactivation (Infections and infestations) | 1 | 0 | 0
Infections, other: bacillus positive blood culture (Infections and infestations) | 1 | 0 | 0
Infection, other- BK positive urine (Infections and infestations) | 1 | 0 | 0
Infections, other; Adenovirus PCR+ (Infections and infestations) | 1 | 0 | 0
Infections, other; RSV+ (Infections and infestations) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
PTT Prolonged (Blood and lymphatic system disorders) | 2 | 0 | 0
Skin, other- Drug reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Vasovagal Reaction (Nervous system disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT02641236/Prot_SAP_000.pdf